CLINICAL TRIAL: NCT02999516
Title: Complex Motor Learning With Motor Imaginary
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Universitario La Salle (Other)
Responsible Party: Principal Investigator, Daniel Muñoz-Garcia, PhD, Centro Universitario La Salle
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: CULaSalle
Record Dates: First submitted 2016-11-24; First posted 2016-12-21 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Learning Disturbance
MeSH Terms: conditions — Learning Disabilities | interventions — Transcranial Direct Current Stimulation; Neurofeedback

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Motor imaginary (Experimental): Intervention with Motor imaginary with video
  Interventions: Other: Motor imaginary
- Non Motor imaginary (Experimental): Intervention with Rest without motor imaginary
  Interventions: Other: Non Motor imaginary
- tDCS (Experimental): tDCS stimulation during 20 minutes in the motor cortex.
  Interventions: Other: tDCS
- tDCS sham (Sham Comparator): tDCS stimulation during 30 seconds in the motor cortex and then 19 minutes and 30 seconds without any stimulation.
  Interventions: Other: tDCS sham
- Neurofeedback (Experimental): EEG monitoring in real time with positive feedback in the computer screen when participants motor cortex is activated.
  Interventions: Other: Neurofeedback
- Neurofeedback sham (Sham Comparator): EEG monitoring in real time with randomized feedback in the computer screen despite the motor cortex activation.
  Interventions: Other: Neurofeedback sham

INTERVENTIONS:
Other: Motor imaginary — Participants imagine doing a motor task watching a video recording
  Arms: Motor imaginary
Other: Non Motor imaginary — Participants watch a television documentary
  Arms: Non Motor imaginary
Other: tDCS — transcranial direct current stimulation (tDCS) stimulation during 20 minutes in the motor cortex (bilaterally) at 1mA of intensity.
  Arms: tDCS
Other: tDCS sham — tDCS stimulation during 30 seconds in the motor cortex (bilaterally) at 1mA of intensity and then 19 minutes and 30 seconds without any stimulation.
  Arms: tDCS sham
Other: Neurofeedback — EEG monitoring of the cerebral cortex in real time with positive feedback in the computer screen when participants motor cortex is activated. The positive feedback consist in an object that moves to the top of the screen when activation occurs in the motor cortex. This task last during 20 minutes.
  Arms: Neurofeedback
Other: Neurofeedback sham — EEG monitoring of the cerebral cortex in real time with randomized feedback in the computer screen despite motor cortex activation. The positive feedback consist in an object that moves to the top of the screen in a randomized time. This task last during 20 minutes.
  Arms: Neurofeedback sham

SUMMARY:
Subjects participate in a motor learning training with a special bicycle. The experimental group proceed with 15 minutes of physical training with the bicycle and 15 minutes of rest where they use motor imaginary. The control group proceed equal except for the motor imaginary intervention.

DETAILED DESCRIPTION:
Subjects participate in a motor learning training with a special bicycle. The experimental group proceed with 15 minutes of physical training with the bicycle and 15 minutes of rest where they use motor imaginary. The control group proceed equal except for the motor imaginary intervention.

Participants will be controlled for vestibular system previous participation.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 29 years old
* Asymptomatic

Exclusion Criteria:

* Subjects with pain
* In medical treatment
* Diagnosed of any disease

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-06 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Time | immediately during the intervention
  Minutes of time when the task is learned

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Superior de Estudios Universitarios La Salle, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Serrano JI, Munoz-Garcia D, Ferrer-Pena R, D'eudeville V, Brero M, Boisson M, Del Castillo MD. Prior cortical activity differences during an action observation plus motor imagery task related to motor adaptation performance of a coordinated multi-limb complex task. Cogn Neurodyn. 2020 Dec;14(6):769-779. doi: 10.1007/s11571-020-09633-2. Epub 2020 Sep 10. PMID 33101530